CLINICAL TRIAL: NCT03342170
Title: Influence of ABO Blood Group on the Risk of Complications in Alcoholic or Viral C Cirrhosis? Analysis From Two French Prospectives National Cohorts CIRRAL and CIRVIR of Patients With Alcoholic or Viral Cirrhosis Child Pugh A
Brief Title: Influence of ABO Blood Group on the Risk of Complications in Alcoholic or Viral C Cirrhosis?
Acronym: ABOCIRRALVIR
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Collaborators: Thong DAO (Unknown); Annie BOREL-DERLON (Unknown); Nathalie GANNE-CARRIE (Unknown); Pierre NAHON (Unknown); Sylvie CHEVRET (Unknown)
Responsible Party: Sponsor
Other Study IDs: ABOCIRRALVIR
Record Dates: First submitted 2017-11-10; First posted 2017-11-14 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2019-08

CONDITIONS: Alcoholic or Viral C Compensated Cirrhosis
MeSH Terms: interventions — Factor V

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — G20210A prothrombin gene mutation Factor 5 Leiden mutation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CIRRAL: alcoholic cirrhosis
  Interventions: Genetic: G20210A prothrombin gene mutation and Factor 5 Leiden mutation
- CIRVIR: Viral cirrhosis
  Interventions: Genetic: G20210A prothrombin gene mutation and Factor 5 Leiden mutation

INTERVENTIONS:
Genetic: G20210A prothrombin gene mutation and Factor 5 Leiden mutation — blood sample

SUMMARY:
The non-O blood group is a risk factor of deep vein thrombosis and recurrence of thromboembolic events, especially when associated with Factor 5 Leiden or prothrombin G20210A mutations. A recent study suggests that non-O blood group may promote portal vein thrombosis in non cirrhotic patients.

In addition, in general population and chronic hepatitis C, non-O blood group combined with one or the other of the above genetic abnormalities is associated with an increased risk of liver fibrosis and accelerated fibrogenesis. The suspected mechanism could be an increased procoagulant factor VIII and an increased Willebrand plasma level, due to a low ADAMTS 13 activity, the result of which is an hypercoagulable state and a microthrombotic process.

In cirrhotic patients procoagulant factors and ADAMTS 13 which are respectively increased and decreased, have be shown to be prognostic markers of hepatocellular function and portal hypertension. It has been hypothesized that the hypercoagulable state and the microthrombotic process could contribute to the worsening of the disease and enoxaparin has been shown to positively modify the prognosis of cirrhosis.

The role of non-O blood group in decompensation of cirrhosis and occurrence of complications including non-tumor portal vein thrombosis has never been studied. The investigators plan a longitudinal observational study to determine the incidence of complications in alcoholic and viral cirrhosis in case of non-O blood group compared to O blood group. The aim of this study is to determine whether ABO blood group may promote complications in alcoholic or viral cirrhosis. This is an ancillary study of two national cohorts assessing natural history and hepatocellular carcinoma risk factors in alcoholic (CIRRAL) and viral (CIRVIR) cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient with either alcoholic or viral C cirrhosis included in national cohorts CIRRAL and CIRVIR

Exclusion Criteria:

* Those of CIRRAL and CIRVIR with None Tumoral Portal Thrombosis prior history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cohorts of cirrhotics patients Child Pugh A followed prospectively to study the natural history of cirrhosis and HCC risk
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-22 (Actual)

PRIMARY OUTCOMES:
cumulated incidence of complications at 3 years | from inclusion to 3 years
  patient follow up during 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle OLLIVIER, MD, Principal Investigator — University Hospital, Caen
Locations (1):
- CHU de CAEN, Caen, France

REFERENCES:
- [Derived] Ollivier-Hourmand I, Repesse Y, Nahon P, Chaffaut C, Dao T, Nguyen TTN, Marcellin P, Roulot D, De Ledinghen V, Pol S, Guyader D, Archambeaud I, Zoulim F, Oberti F, Tran A, Bronowicki JP, D'Alteroche L, Ouzan D, Peron JM, Zarski JP, Bourliere M, Larrey D, Louvet A, Cales P, Abergel A, Mathurin P, Mallat A, Blanc JF, Nguyen-Khac E, Riachi G, Alric L, Serfaty L, Antonini T, Moreno C, Attali P, Thabut D, Pilette C, Grange JD, Silvain C, Carbonell N, Bernard-Chabert B, Goria O, Wartelle C, Moirand R, Christidis C, Perlemuter G, Ozenne V, Henrion J, Hillaire S, Di Martino V, Amiot X, Sutton A, Barget N, Chevret S, Ganne-Carrie N; ANRS CO12 CIRVIR, CIRRAL groups. ABO blood group does not influence Child-Pugh A cirrhosis outcome: An observational study from CIRRAL and ANRS CO12 CIRVIR cohorts. Liver Int. 2022 Jun;42(6):1386-1400. doi: 10.1111/liv.15159. Epub 2022 Jan 17. PMID 35025128